CLINICAL TRIAL: NCT01123512
Title: The Kiva® System as a Vertebral Augmentation Treatment - A Safety and Effectiveness Trial
Brief Title: The Kiva® System as a Vertebral Augmentation Treatment
Acronym: KAST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Benvenue Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BEN005
Record Dates: First submitted 2010-05-11; First posted 2010-05-14 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Spinal Fractures; Fractures, Compression; Back Injuries
Keywords: Vertebral Compression Fracture; Kyphoplasty; Spine; Vertebral Body Compression Fracture; Back Pain
MeSH Terms: conditions — Spinal Fractures; Fractures, Compression; Back Injuries; Back Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kiva VCF Treatment System (Experimental)
  Interventions: Device: Vertebral augmentation
- Balloon Kyphoplasty (Active Comparator)
  Interventions: Device: Vertebral augmentation

INTERVENTIONS:
Device: Vertebral augmentation — Vertebral augmentation for one or two osteoporotic vertebral compression fractures

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the Kiva VCF Treatment system in comparison to balloon kyphoplasty for the treatment of osteoporotic vertebral compression fractures of the thoracic or lumbar spine.

ELIGIBILITY:
Inclusion Criteria

Patients must meet all of the following inclusion criteria below to be included as research subjects:

1. The patient is at least 50 years of age
2. The patient has a score on the back pain visual analog scale (VAS) of ≥70 mm after 2 to 6 weeks of conservative care OR a VAS of ≥ 50 mm after 6 weeks of conservative care
3. The patient has an Oswestry Disability Index (ODI) score of ≥ 30%
4. The patient has radiographic evidence of one or two (1-2) A 1.1, A 1.2, A 1.3. fractures as classified by the AO Spine Fracture classification, due to primary or secondary osteoporosis in the thoracic and / or lumbar spine. Note that patients are eligible if they have had treatment of or healed VCF(s) at any non-index level
5. The patient has central pain over the spinous process(es) upon palpation at the Index level(s)
6. The Index fracture(s) is / are acute or persistent (not healed), as demonstrated by T2 weighted STIR MRI (or bone scan if patient is contraindicated for MRI
7. The Index fracture(s) has / have failed conservative care of at least 2 weeks but no longer than 6 months
8. The Index fracture(s) shows radiographic evidence of at least 5% vertebral collapse
9. The pedicle identified for access to the index fracture has a diameter that is ≥ 6 mm
10. The patient is mentally capable and willing to sign a study-specific informed consent as documentation of the informed consent process prior to any study procedures
11. The patient is willing and able to comply with all study requirements including follow-up visits and radiographic assessments

Exclusion Criteria

Patients will not be allowed to participate in the study if they meet any of the exclusion criteria below:

1. The index fracture(s) has/have been caused by high-energy trauma
2. The index fracture(s) has / have known tumor involvement
3. The index fracture(s) is/are diagnosed as an osteonecrotic fracture(s) by the treating physician
4. The Index fracture(s) is a/are translational force fracture(s) (A2.1, 2.2, 2.3)
5. The index fracture(s) is a/are burst fracture(s) (A 3.3., B or C type) or pedicle fracture(s) with posterior cortical wall disruption
6. The index fracture(s) has / have posterior vertebral wall displacement occupying more than 20% of the cross sectional area of the spinal canal
7. The index fracture(s) has / have severe deformity with reduction of >75% in any height and accompanying area, using adjacent level as comparison
8. The index level(s) has / have undergone previous surgical treatment for a vertebral body compression fracture or other surgical procedure at the index level(s)
9. Angulation of index fracture(s) makes treatment with Kiva System impossible (at discretion of surgeon)
10. The pedicle identified for access to the index fracture has a diameter less than 6 mm
11. The patient has Paget's disease
12. The patient has a BMI > 35
13. The patient has uncontrolled diabetes as characterized by hemoglobin HbA1c >7% and/or blood sugar >180mg/dL
14. The patient has severe cardiopulmonary deficiencies
15. The patient has myelopathy
16. The patient is on long-term steroid therapy (steroid dose ≥ 30 mg /day for > 3 months)
17. A medical contraindication to spinal surgery and/or general anesthesia, such as coagulopathy (with a threshold for normal being INR ≤ 1.5, PTT within lab normal range, and platelet count > 100,000)
18. The patient has spinal canal compromise causing clinical manifestations of cord, neural foramen, or nerve root compression at the level(s) to be treated;
19. The patient has neurologic symptoms or deficits or radiculopathy related to the VCF
20. The patient has pain based on clinical diagnosis of herniated nucleus palposus or severe spinal stenosis (progressive weakness or paralysis)
21. The patient has indications of instability related to the index fracture (≥ 30 degrees of kyphosis, translation >4mm, interspinous process widening, > Grade 1 spondylolisthesis and/or > 25 degrees of scoliosis if the index level is included in the curve)
22. The patient has planned spine surgery for any disorder during or up to 30 days after the study treatment
23. The patient has had spine surgery for any disorder in the 30 days prior to enrollment
24. The patient has a documented active systemic or local infection, such as osteomyelitis or discitis, with a WBC > 15.0 x 10^3/µL and a temperature > 101.5°F
25. The patient has a known allergy to the investigational device materials and / or acrylics / polymethylmethacrylate (PMMA) or a hypersensitivity to monomers
26. The patient has been diagnosed with hemorrhagic diathesis
27. The patient has uncontrolled psychiatric illness or severe dementia
28. The patient has a baseline back pain visual analog scale (VAS) of <50 mm if patient has at least 6 weeks of conservative care or <70 mm if patient has 2-6 weeks conservative care
29. The patient has a baseline Oswestry Disability Index (ODI) score of <30%
30. The patient is currently on anti-cancer therapy or anti-HIV therapy
31. Patient has autoimmune or inflammatory rheumatic disease
32. Patient's life expectancy is less than the study duration or undergoing palliative care
33. The patient is known to be a current alcohol or drug abuser
34. The patient is known to be involved in medical litigation including Workmen's Compensation
35. The patient is a prisoner
36. The patient is participating in another investigational study that has a potential for effect to the study treatment or the study endpoints
37. The patient is pregnant or considering getting pregnant during study participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2010-07; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven R. Garfin, MD, Principal Investigator — University of California, San Diego, CA; Sean M. Tutton, MD, FSIR, Principal Investigator — Medical College of Wisconsin
Locations (21):
- United States (15):
  - CORE Orthopaedic Medical Center, Encinitas, California
  - El Camino Hospital, Mountain View, California
  - Radiological Associates of Sacramento, Sacramento, California
  - St. Mary's Spine Center, San Francisco, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Evanston Hospital, Evanston, Illinois
  - Adventist Hospital, Hinsdale, Illinois
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - Sierra Regional Spine Institute, Reno, Nevada
  - Clinical Radiology of Oklahoma, Edmond, Oklahoma
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- CHC Saint Joseph, Liège, Belgium
- Canada (2):
  - Toronto Western Hospital, Toronto, Ontario
  - Montreal General Hospital, Montreal, Quebec
- CHU Amiens Sud, Amiens, France
- Germany (2):
  - Universitatsklinikum Bonn, Bonn
  - Klinikum Ernst von Bergmann gGmbH, Potsdam

REFERENCES:
- [Derived] Beall DP, Coe JD, McIlduff M, Bloch D, Hornberger J, Warner C, Tutton S. Serious Adverse Events Associated with Readmission Through One Year After Vertebral Augmentation with Either a Polyetheretherketone Implant or Balloon Kyphoplasty. Pain Physician. 2017 Sep;20(6):521-528. PMID 28934783

RESULTS

PARTICIPANT FLOW:
Groups:
- Kiva VCF Treatment System: The Kiva® VCF Treatment System is a multi-component, single-use device designed for obtaining unilateral access to the vertebral body in order to deliver the Kiva Implant and bone cement to stabilize osteoporotic vertebral fractures. The Kiva procedure involved placement of the Kiva Implant into the vertebral body followed by injection of PMMA into the Kiva Implant.
- Balloon Kyphoplasty: The balloon kyphoplasty procedure involved placing an inflatable bone tamp into the vertebral body that was then inflated under fluoroscopic guidance to create a void. This void was then filled with PMMA.
Period: Overall Study
Arm/Group | Kiva VCF Treatment System | Balloon Kyphoplasty
Started | 153 | 147
Completed | 127 | 126
Not Completed | 26 | 21

BASELINE CHARACTERISTICS:
Population: As-Treated population
Groups:
- Total: Total of all reporting groups
Arm/Group | Kiva VCF Treatment System | Balloon Kyphoplasty | Total
Number analyzed (Participants) | 144 | 141 | 285
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.03 (8.82) | 75.09 (9.62) | 75.57 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 211
  Male | 39 | 35 | 74

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Study Success
Description: Patient success will be defined as:
  1. Reduction in VCF fracture-related pain at 12 months by >15 mm from baseline as measured by a 100 mm Visual Analog Scale (VAS),
  2. Maintenance or improvement in function at 12 months from baseline as measured by the 100 point Oswestry Disability Index (ODI), and
  3. Absence of device-related serious adverse events, defined as device-related adverse events requiring surgical reintervention or retreatment at the index level, including revision, removal, reoperation, and/or supplemental fixation
Time Frame: 12 Month Post-op
Measure: Number; unit: participants
Arm/Group | Kiva VCF Treatment System | Balloon Kyphoplasty
Number analyzed (Participants) | 127 | 126
participants | 120 | 123
Statistical Analysis 1: Comparison: Kiva VCF Treatment System vs Balloon Kyphoplasty; Test type: Non-Inferiority or Equivalence — Pr( Pt - Pc > -12.5% | data), calculated using Bayesian multiple imputation for missing 12-month values, as specified in the protocol. The Kiva System is declared non-inferior to control if Pr( Pt - Pc > -12.5% | data)> 96.6%; Bayesian test of proportions — Pr( Pt - Pc > -12.5% | data), calculated using Bayesian multiple imputation for missing 12-month values, as specified in the protocol. The Kiva System is declared non-inferior to control if Pr( Pt - Pc > -12.5% | data)> 96.6%; % Probability of Equivalence = 99.92 = 99.92

ADVERSE EVENTS:
Arm/Group | Kiva VCF Treatment System | Balloon Kyphoplasty
Serious Adverse Events (participants affected / at risk) | 44/153 | 51/147
Other Adverse Events (participants affected / at risk) | 81/153 | 80/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kiva VCF Treatment System (N=153) | Balloon Kyphoplasty (N=147)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Plasmacytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Spleen disorder (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 2 (4)
Dizziness (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 3 (3)
Unstable angina (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal functional disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mesenteric artery embolism (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 2 (2) | 1 (2)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus colitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Peridiverticulitis (Infections and infestations) | 1 (2) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (2) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 4 (4)
Airway complication of anesthesia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Muscle injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 10 (14) | 13 (20)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Spondylolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Lung cancer metas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Myelodysplastics (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Spinal menigioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Myasthenia gravis (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1)
Fear of falling (Psychiatric disorders) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 1 (1) | 0 (0)
Pseudodementia (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 2 (2) | 0 (0)
renal disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Bladder catheter replacement (Surgical and medical procedures) | 0 (0) | 1 (1)
Drug delivery device implantation (Surgical and medical procedures) | 1 (1) | 0 (0)
Subdural haematoma evacuation (Surgical and medical procedures) | 0 (0) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (2)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kiva VCF Treatment System (N=153) | Balloon Kyphoplasty (N=147)
Oedema peripheral (General disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 1 (1) | 3 (3)
Herpes zoster (Infections and infestations) | 3 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (4)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Spinal compression fracture (Injury, poisoning and procedural complications) | 49 (74) | 40 (58)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 39 (52) | 41 (45)
Motor dysfunction (Nervous system disorders) | 0 (0) | 3 (3)
Reflexes abnormal (Nervous system disorders) | 7 (8) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No